CLINICAL TRIAL: NCT04283409
Title: Which Exercise for Low Back Pain? Predicting Response to Exercise Treatments for Patients With Low Back Pain - a Validation Randomized Controlled Trial
Brief Title: Which Exercise for Low Back Pain? Predicting Response to Exercise for Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Macquarie University, Australia (Other); Laval University (Other); The University of Queensland (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Luciana Macedo, Associate Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HiREB#7986
Record Dates: First submitted 2020-01-24; First posted 2020-02-25 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Non-specific Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Given the exercise nature of the study it is not possible to blind therapists or patients, however; assessors will remain blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Control Exercise (Experimental): The primary goal of motor control exercises is to retrain optimal control and coordination of the spine. It uses principles of motor learning such as segmentation, simplification and task-specific practice to retrain control of trunk muscles activation, alignment and movement. The first stage of the treatment involves assessment of the postures, movement patterns and muscle activation associated with symptoms and a retraining program designed to improve activity of muscles assessed to have poor control (usually the deep trunk muscles). Participants are taught how to contract these muscles independently. During this stage additional exercises for breathing control, posture of spine and movement are performed. The second stage of the treatment involves the progression of the exercises towards functional activities, firstly using static then dynamic tasks. Education is also included.
  Interventions: Other: Motor Control Exercises
- Graded Activity (Experimental): The primary goal of graded activity is to address individual modifiable contextual factors associated with the pain experience such as self-efficacy, pain-related fear, kinesiophobia and unhelpful beliefs/behaviors about back pain while at the same time addressing physical impairments such as endurance, muscle strength and balance. A primary goal of the program is to increase activity tolerance by performing individualized and submaximal exercises in addition to ignoring illness behaviors and reinforcing well behaviors. Activities in the program are progressed in a time-contingent manner from the baseline assessed ability to a target goal set jointly by patient and therapist. Cognitive-behavioral principles are used to help patients overcome the natural anxiety associated with pain and activities.
  Interventions: Other: Graded activity

INTERVENTIONS:
Other: Graded activity — Exercise therapy using principles of cognitive behavioral therapy and education
  Arms: Graded Activity
Other: Motor Control Exercises — Exercise therapy using principles of motor control and motor learning and education
  Arms: Motor Control Exercise

SUMMARY:
Exercise therapy is the most recommended treatment for chronic low back pain. There is a wide range of exercises available and research studies have shown that no exercise is superior to another. The problem is that the effects of exercise in reducing pain and disability are small to moderate. Researchers and clinicians believe that different patients may best respond to different types of exercises. This means that if patients could be better matched to specific exercises, then the effects of exercise would be greater. A study conducted by the investigators of this study tested whether patient's characteristics could predict outcomes to two of the most common exercises for low back pain: motor control exercises or graded activity. The results showed that a simple questionnaire (Lumbar Spine Instability Questionnaire) could identify patients who responded best to either exercise. Patients with low clinical instability (measured by the questionnaire) responded best to graded activity. Patients with high clinical instability responded best to motor control exercises.These results were the first to show that better matching patients to specific exercises improves outcomes. Although these results have the potential to significantly improve the delivery of exercises for low back pain, validation of the results in a high-quality study with a large group of patients is a prerequisite to clinical implementation. The aim of this study is to conduct a randomized controlled trial comparing the effects of graded activity to motor control exercises and identify groups of respondents to these exercises. The study will also include the evaluation the costs and benefits of these interventions and the potential impact of matched treatment to patients and the health care system. The results of this study has the potential to increase the effects of exercise in low back pain and consequently lead to better patient outcomes and decreased health related costs.

DETAILED DESCRIPTION:
Background:

Clinical practice guidelines consistently endorse exercise therapy for the treatment of low back pain (LBP). While exercise is more effective than no intervention, the effect size of exercise, like other treatments for LBP, is relatively small. While there are many forms of exercise therapies available (e.g. general exercise, pilates), there is no clear evidence of superiority of one exercise over another. A widely held belief is that the small effect for exercise is due to the heterogeneity of people presenting with LBP and if individual patients could be better matched to the optimal types of exercise, then the effects of treatment would be greater.A recently published study conducted by the study investigators provided preliminary evidence supporting the hypothesis of better outcomes when patients are matched to the appropriate exercise. The study demonstrated that a simple 15-item questionnaire, the Lumbar Spine Instability Questionnaire (LSIQ), could identify patients who responded best to either of the most common exercise approaches for LBP. Participants who had low scores on the LSIQ had better outcomes with graded activity while those with higher scores had better outcomes with motor control exercise. Theoretically, motor control would work best on those that have poor coordination and control of the trunk muscles and graded activity would work best on those with unhelpful beliefs and attitudes towards back pain. Although the results of this study have the potential to transform exercise treatment for LBP, validation and confirmation off the results in a fully powered study using an independent sample is essential before recommending implementation in clinical practice. Validation and impact analysis are crucial steps in the investigation of effect modification models.

Research aims:

The primary aim of this study is to evaluate whether pre-identified baseline characteristics, including the LSIQ, can modify the response to two of the most prominent exercise therapies (graded activity and motor control) for non-specific LBP.

The secondary aims include a cost-effectiveness analysis of a potential stratified care model.

Exploratory aims include the evaluation of potential new effect modifiers that may strengthen the initial prediction model. This include measures of central pain mechanisms to differentiate nociceptive, neuropathic and nociplastic pain.

Methods:

Participants (414) will be recruited by primary care professionals and will be randomized (1:1) to receive either motor control exercises or graded activity. Participants will receive 12 sessions of exercise therapy,delivered by a physiotherapist, over an 8-week period. The primary outcome will be disability at 2 months measured using the Oswestry Disability Index. Secondary outcomes will be pain, function and quality of life measured at 2, 6 and 12 months.

Potential effect modifiers will be the LSIQ, self-efficacy, coping strategies, kinesiophobia and measures of nociceptive pain and central sensitization. The study will follow specific guidelines for the conduction of effect modification studies.

Expected outcomes:

The results of this study will provide the foundation for the implementation of the study results in large scale which would significantly improve the effects of exercise for LBP. Furthermore, it will provide cost-effectiveness information to guide clinical decision making. Implementation of this approach would be simple as both treatments are already widely used and the method to identify subgroups of responders to each approach is straight forward, quick and at no cost.

ELIGIBILITY:
Inclusion Criteria:

* chronic non-specific LBP (>3 months) with or without leg pain
* back pain being the primary musculoskeletal complaint of the patient
* between 18 to 80 years of age,
* English speaking (to allow response to questionnaires and communication with physiotherapist),
* moderate or greater pain or disability measured using question 7 and 8 of the SF-36,34
* moderate or high risk classification on the STarT Back Tool indicating appropriateness of physiotherapy and thus an exercise program.

Exclusion Criteria:

* nerve root compromise (2 strength, reflex or sensation affected for the same nerve root)
* suspected or confirmed serious pathology (e.g. infection, fracture, cancer, inflammatory arthritis, cauda equina syndrome)
* pregnancy
* scheduled or on the wait list for surgery during trial period
* cognitive impairment that precludes participant from completing study questionnaires or comply with exercise recommendations (e.g. dementia, Alzheimers)
* severe neuromuscular condition (e.g. spinal cord injury) that precludes participant from engaging in activity exercise.
* clinical assessment indicating that the participant is not suitable for active exercises (by a family physician, or using the Physical Activity Readiness Questionnaire).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 2 months
  disease specific disability questionnaire; total score from 0-100 (higher scores represent worse disability)

SECONDARY OUTCOMES:
Patient Specific Functional Scale | 0, 2, 6 and 12 months
  Rate 3 problematic activities; average of the 3 activities generate a total score from 0-10 (lower scores represent worse function)
Pain Numeric Ranting Scale | 0, 2, 6 and 12 months
  Pain over the last week; total score from 0-10 (higher scores represent worse pain)
EQ-5D-5L | 0, 2, 6 and 12 months
  Health related quality of life; index score form 0-100 (lower scores represent lower quality of life) in addition Quality- Adjusted Life Years QUALYS) will be calculated.
IMPACT of low back pain - PROMIS-9 | 0, 2, 6 and 12 months
  NIH recommended IMpACT: pain intensity, pain interference and functional status; scored from 8-50 (higher score represents more pain impact)

OTHER OUTCOMES:
Lumbar Spine Instability Questionnaire: Effect Modifier: | 0, 2 and 12 months
  Measure self reported 'clinical instability'; total score 0-15 (higher scores represent more instability) (Participants will be dichotomized as having instability >=9 or no instability <9)
Effect Modifier: OREBRO LBP screening questionnaire | 0, 2 and 12 months
  Measures attitudes and behavior towards pain; total score 11-192 (higher scores represent worse attitudes and behavior) (Median scores will be used to dichotomize participants into high and low scores)
Effect Modifier: TAMPA scale of kinesiophobia | 0, 2 and 12 months
  Measures fear of movement; total score from 0-52 (higher scores represent worse kinesiophobia) (median scores will be used to dichotomize participants into high or low scores)
Effect Modifier: Coping strategies questionnaire | 0, 2 and 12 months
  Measures coping strategies; total score from 0-36 (higher scores represent worse coping) (median scores will be used to dichotomize participants into high or low scores)
Effect Modifier: painDetect Questionnaire | 0, 2 and 12 months
  This questionnaire total score >18 will classify participants into neuropathic or non neuropathic pain(dichotomous outcome)
Effect Modifier: SMART clinical checklist | 0, 2 and 12 months
  The sub-cores of the questionnaire as per SMART et al will be used to used to discriminate between nociceptive, neuropathic and nociplastic pain. (Nominal scale)
Effect Modifier: Pain Pressure Threshold Assessment | 0, 2 and 12 months
  PPT will be assessed at the lumbar spine (point with most pain) and thumbnail (distal point) using an algometer. Difference in PPT between local and distal sites will be included in the analysis. (high scores will represent more nociplastic pain)
Publicly funded health care costs | 1 year prior to intervention, 12 months follow-up
  Health care utilization costs will be extracted from the Ontario Health Funder database and an IC/ES (Institute for Clinical Evaluative Sciences) algorithm will be used to calculate health care utilization dollars per participant.
Patient direct health care costs | 12 months follow-up
  Direct health care costs (e.g. physiotherapy, travel) will be calculated following the completion of a health care utilization questionnaire. Total utilization will be reported as dollars per participants
Societal health care costs | 12 months follow-up
  Indirect health care costs (e.g. work lost productivity) will be calculated following the completion of a health care utilization questionnaire. Total utilization will be reported as dollars per participants

CONTACTS AND LOCATIONS:
Overall Officials: Luciana G Macedo, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data may be requested directly to the principal investigator or may be made available upon publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available following publication of the results.
Access Criteria: Ethics approval will be required for any secondary analysis of data as per HiREB approval.

REFERENCES:
- [Background] Macedo LG, Maher CG, Hancock MJ, Kamper SJ, McAuley JH, Stanton TR, Stafford R, Hodges PW. Predicting response to motor control exercises and graded activity for patients with low back pain: preplanned secondary analysis of a randomized controlled trial. Phys Ther. 2014 Nov;94(11):1543-54. doi: 10.2522/ptj.20140014. Epub 2014 Jul 10. PMID 25013000
- [Derived] Macedo LG, Hodges PW, Bostick G, Hancock M, Laberge M, Hanna S, Spadoni G, Gross A, Schneider J. Which Exercise for Low Back Pain? (WELBack) trial predicting response to exercise treatments for patients with low back pain: a validation randomised controlled trial protocol. BMJ Open. 2021 Jan 20;11(1):e042792. doi: 10.1136/bmjopen-2020-042792. PMID 33472786